CLINICAL TRIAL: NCT04831684
Title: Effects of a Novel mGluR5 Negative Allosteric Modulator on Alcohol Drinking, Neurochemistry, and Brain Reactivity to Alcohol Cues in Alcohol Use Disorder
Brief Title: Novel mGluR5 Modulator Effects on Alcohol Drinking and MRI Outcomes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, James Prisciandaro, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Pro00102334
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator)
  Interventions: Drug: Placebo
- Group B (Experimental)
  Interventions: Drug: GET73

INTERVENTIONS:
Drug: Placebo — Participants will be getting placebo for 8 days of dosing.
  Arms: Group A
Drug: GET73 — Participants will be getting GET73 for 8 days of dosing.
  Arms: Group B

SUMMARY:
This study evaluates the effects of the medication GET73 among non-treatment-seeking individuals who regularly drink alcohol. Participants in the study will take GET73 or placebo for an 8-day study. There are 4 study visits including 2 MRI scans.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-40 (to focus on an age group still on a trajectory of increasing alcohol consumption, consistent with our pilot data and past iterations of the ARC).
2. Meets Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for current Alcohol Use Disorder, with at least Moderate severity.
3. Reports drinking, on average, at least 20 standard alcoholic drinks per week for at least the past 3 months.
4. Currently not engaged in, and does not want treatment for, alcohol-related problems.
5. Able to read and understand questionnaires and informed consent.
6. Lives within 50 miles of the study site.
7. Able to maintain abstinence from alcohol the evening prior to appointments (without the aid of detoxification medications), as determined by self-report and breathalyzer measurements.
8. Amenable to drinking liquor in fruit juice.

Exclusion Criteria:

1. Current DSM-5 diagnosis of any other substance use disorder except Nicotine Use Disorder.
2. Any psychoactive substance use (except marijuana and nicotine) within the last 30 days, as indicated by self-report and urine drug screen. For marijuana, no use within the last seven days by verbal report and negative (or decreasing) urine THC levels.
3. Current DSM-5 Axis I diagnosis, including major depression, panic disorder, obsessive-compulsive disorder, post-traumatic stress disorder, bipolar affective disorder, schizophrenia, dissociative disorders, eating disorders, or any other psychotic or organic mental disorder.
4. Current suicidal ideation or homicidal ideation.
5. Using CYP2C19 and/or CYP3A4 inhibitors or inducers in the 14 days before dosing or during the study.
6. Need for maintenance or acute treatment with any psychoactive medication, including antiepileptic medications.
7. Currently taking medication known to affect alcohol intake (e.g., disulfiram, naltrexone, acamprosate, topiramate).
8. History of severe alcohol withdrawal (e.g., tremor, sweating, anxiety, seizure, delirium tremens), as evidenced by self-report and assessment with Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar).
9. Clinically significant medical problems such as cardiovascular, renal, gastrointestinal, or endocrine problems that would impair participation or limit medication ingestion.
10. Past alcohol-related medical illness, such as gastrointestinal bleeding, pancreatitis, or peptic ulcer.
11. Has hepatocellular disease indicated by elevations of SGPT (ALT) or SGOT (AST) greater than 2.5 times normal at screening.
12. Females of childbearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
13. Current charges pending for a violent crime (not including DUI-related offenses).
14. Lack of a stable living situation.
15. Presence of ferrous metal in the body, as evidenced by metal screening and self-report.
16. Severe claustrophobia or extreme obesity that preclude placement in the MRI scanner.
17. Neurological disease or history of head injury with > 2 minutes of unconsciousness.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Number of drinks consumed during bar-lab paradigm (free drinking period) | 165 minutes
Change in Gamma aminobutyric acid (GABA) and glutamate levels | baseline to day 7
  Acquired via spectroscopy sequence completed at baseline and day 7 scans
Levels of cortical activation to visual cues of alcohol | baseline to day 7
  Acquired via functional magnetic resonance imaging completed at baseline and day 7 scans

CONTACTS AND LOCATIONS:
Overall Officials: James Prisciandaro, Principal Investigator — Medical University of South Carolina
Locations (1):
- Charleston Alcohol Research Center, Institute of Psychiatry, Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Per NOT-AA-19-020, this study will submit and share data with NIAAA Data Archive, a data repository housed within the NIMH Data Archive. This includes broad sharing of all research subjects' de-identified data.
Supporting Information: Study Protocol
Time Frame: De-identified participant data will be uploaded to the NIMH Data Archive twice yearly (by April 1 and October 1) during the course of this study, and will remain available with no end date.
Access Criteria: Data and supporting documentation submitted to the NIMH Data Archive may be accessed and used broadly by approved users for research and other activities as authorized by and consistent with law.
URL: https://nda.nih.gov/niaaa/award/data-sharing-expectations.html

DOCUMENTS (1):
  • Informed Consent Form (2025-09-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT04831684/ICF_000.pdf